CLINICAL TRIAL: NCT03951948
Title: Optimys Femoral Stem for Total Hip Replacement - a Clinical and Radiologic Follow-up of Minimum One Year
Brief Title: Optimys Femoral Stem for Total Hip Replacement
Acronym: Optihip
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00563; ch19Saxer
Record Dates: First submitted 2019-05-06; First posted 2019-05-16 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Short Stem Prosthesis; Optimys Femoral Stem
Keywords: total hip replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective analysis of surgical performance, clinical and radiologic outcome — retrospective analysis of surgical performance, clinical and radiologic outcome

SUMMARY:
This retrospective observational study analyses the surgical performance, clinical and radiologic outcome as well as the rate of infections with a main focus on revision surgeries after primary implantation of the Optimys short stem femoral prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with an Optimys femoral component at the University Hospital Basel between 29.10.2013 and 29.10.2018

Exclusion Criteria:

* Clinical follow up at another Institution
* Documented dissent in study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a proximal femoral fracture at the University Hospital Basel between 29.10.2013 (date of introduction of the Optimys femoral component at the university hospital Basel) and 29.10.2018.
Sampling Method: Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
rate of reoperations | one year follow-up period after Optimys femoral stem surgery
  rate of reoperations after primary implantation of the Optimys short stem prosthesis

SECONDARY OUTCOMES:
rate of cortical hypertrophy | at one year follow-up after Optimys femoral stem surgery
  rate of cortical hypertrophy
rate of fractures | one year follow-up period after Optimys femoral stem surgery
  rate of fractures after the implantation of short stem femoral implants
rate of infections | one year follow-up period after Optimys femoral stem surgery
  rate of infections after the implantation of short stem femoral implants
anatomic alignment on anterior-posterior (ap) view in Degree° | at one year follow-up after Optimys femoral stem surgery
  radiologic outcome defined by preciseness of the anatomic alignment compared to the contralateral side
subsidence | at one year follow-up after Optimys femoral stem surgery
  radiologic outcome defined by rate of subsidence after the implantation of short stem femoral implants (mm)
pain at rest (yes/no) | at one year follow-up after Optimys femoral stem surgery
  clinical outcome defined by pain at rest (yes/no)
pain under stress (yes/no) | at one year follow-up after Optimys femoral stem surgery
  clinical outcome defined by pain under stress (yes/no)
use of analgetics (yes/no) | at one year follow-up after Optimys femoral stem surgery
  clinical outcome defined by use of analgetics (yes/no)
use of walking aids | at one year follow-up after Optimys femoral stem surgery
  clinical outcome defined by use of walking aids
extent of periarticular ossification (PAO) according to Brooker classification system | at one year follow-up after Optimys femoral stem surgery
  Brooker classification system divides severity of PAO into 4 types:
  A: islands of bone within the soft tissues about the hip B: bone spurs originating from the pelvis or proximal end of the femur, leaving at least 1 cm between opposing bone surfaces C: bone spurs originating from the pelvis or proximal end of the femur, reducing the space between opposing bone surfaces to less than 1 cm D: bone ankylosis of the hip

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clauss, Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland